CLINICAL TRIAL: NCT01871740
Title: Enalapril Maleate and Folic Acid Tablets for Prevention of Chronic Kidney Diseases in Patients With Hypertension: a Double-blind Randomized Controlled Trial
Brief Title: CSPPT- Chronic Kidney Diseases Study
Acronym: CSPPT-CKD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor and the PIs both agreed that the CSPPT-CKD should be a sub-study of the CSPPT insted of an independent randomized trial.
Sponsor: Shenzhen Ausa Pharmed Co.,Ltd (Industry)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ausa-CSPPT-CKD
Record Dates: First submitted 2013-05-29; First posted 2013-06-07 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension; Hyperhomocysteinemia
Keywords: Folic acid; Renal function decline; Hypertension; Hyperhomocysteinemia; Chronic kidney disease; MTHFR C677T genotype; Randomized controlled trial
MeSH Terms: conditions — Hypertension; Hyperhomocysteinemia; Renal Insufficiency, Chronic | interventions — Enalapril; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enalapril maleate and folic acid tablets (Experimental): A fixed combination drug is given. The dose is fixed in enalapril 10 mg / folic acid 0.8 mg per day.
  Interventions: Drug: Enalapril maleate and folic acid tablets
- Enalapril maleate (Active Comparator): Enalapril maleate 10 mg per day is given
  Interventions: Drug: Enalapril maleate

INTERVENTIONS:
Drug: Enalapril maleate and folic acid tablets — Enalapril maleate and folic acid tablets, (10mg/0.8mg)/tablet, taken orally and once daily for a maximum of 5 years. Combination with other anti-hypertension drugs are allowed.
  Arms: Enalapril maleate and folic acid tablets
Drug: Enalapril maleate — Enalapril, 10mg/tablet, taken orally once daily for a maximum of 5 consecutive years. Combination with other anti-hypertension drugs are allowed.
  Other Names: Lameiya(Yabao Pharmaceutical)
  Arms: Enalapril maleate

SUMMARY:
The purpose of this trial is to confirm that enalapril maleate and folic acid tablets is more effective in preventing renal function decline among the patients with primary hypertension when compared to enalapril maleate.

DETAILED DESCRIPTION:
Elevated blood concentration of homocysteine (Hcy) has been suggested as a modifiable, independent risk factor for coronary artery disease, stroke, and deep vein thrombosis. Prevalence of hyperhomocysteinemia and folic acid deficiency in China are significantly higher than those in Europe and USA. The investigators' preliminary research demonstrated that blood concentration of Hcy was negatively correlated to estimated glomerular filtration rate (eGFR), a key index of kidney function. However, the question as to whether Hcy-lowering therapy with folic acid can reduce the risk of chronic kidney disease(CKD) remains to be answered.

This study, exploiting the hypertensive population of CSPPT trial (ClinicalTrials.gov register number: NCT00794885), is intended to compare the effects of enalapril maleate and folic acid tablets versus enalapril maleate in preventing renal function decline among the patients with primary hypertension. The results from this trial may have the potential to transform current clinical and public health findings into practice in the prevention of chronic kidney disease(CKD) in China.

ELIGIBILITY:
Inclusion Criteria:

* BP≥140/90 mmHg in both of the two screening visits or currently under anti-hypertension treatment;
* 45-75 years old;
* Successful determination of methylenetetrahydrofolate reductase (MTHFR) C677T genotype;
* For pre-menopausal women, agreed to use contraceptives during the trial;
* Signed the written informed consent.

Exclusion Criteria:

* Having a history of stroke;
* Having a history of myocardial infarction;
* Having a history of physician diagnosed heart failure;
* Post- coronary revascularization;
* Severe somatic disease such as cancer;
* Secondary hypertension;
* Congenital or acquired organic heart diseases;
* Contraindicated to angiotensin-converting enzyme inhibitor (ACEI);
* Having a history of ACEI adverse effects;
* Currently long-term use of folic acid or vitamin B12 or vitamin B6;
* Pregnant or child breastfeeding women;
* Severe mental disorders;
* Lab tests indicating abnormal liver or kidney function;
* Unwilling to participate the trial;
* Unwilling to change the current antihypertensive treatment.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Renal function decline | Serum creatinine was examined at baseline and at the final visit (5 years) of the trial.
  Renal function decline was defined based on one of more of the following :
  (1) A certain drop in eGFR, was defined as a drop in GFR category (≥90[G1], 60-89[G2], 45-59[G3a], 30-44[G3b], 15-29[G4], <15[G5] ml/min/1.73m2) accompanied by a 25% or greater drop in eGFR from baseline; (2) Rapid progression, was defined as a sustained decline in eGFR of more than 5 ml/min/1.73m2/yr.

SECONDARY OUTCOMES:
Average decline rate in eGFR (ml/min/1.73m2/yr). | Serum creatinine was examined at baseline and at the final visit (5 years) of the trial.
New-onset chronic kidney disease based on eGFR（eGFR<60 ml/min/1.73 m2） | Serum creatinine was examined at baseline and at the final visit (5 years) of the trial.
New-onset albuminuria | Albuminuria was examined at baseline and at the final visit (5 years) of the trial.
A composite of renal events. | Every 3 months during the trial, up to 5 years
  The composite endpoint is consisted of: 1)End stage renal disease (ESRD);2)Doubling of serum creatinine; and 3)Renal disease-induced death.

CONTACTS AND LOCATIONS:
Overall Officials: Fanfan Hou, MD, Principal Investigator — Division of Nephrology, Nanfang Hospital, Southern Medical University; Xin Xu, MD, Principal Investigator — Guangdong Provincial Institute of Nephrology
Locations (2):
- China (2):
  - Anqing Branch, Anhui Institute of Biomedical Research, Anqing, Anhui
  - Lianyungang Center for Advanced Research in Cardiovascular Diseases, Lianyungang, Jiangsu